CLINICAL TRIAL: NCT05047536
Title: A Phase 1 Study of KZR-261, a Small Molecule Sec61 Inhibitor, in Subjects With Advanced Solid Malignancies
Brief Title: KZR-261 in Subjects With Advanced Solid Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision.
Sponsor: Kezar Life Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KZR-261-101
Record Dates: First submitted 2021-09-03; First posted 2021-09-17 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Advanced/Metastatic Solid Tumor
Keywords: melanoma; uveal melanoma; colorectal cancer; castration-resistant prostate cancer; mesothelioma
MeSH Terms: conditions — Neoplasm Metastasis; Melanoma; Uveal Melanoma; Colorectal Neoplasms; Mesothelioma | interventions — Injections

STUDY DESIGN:
Intervention Model Description: All participants received 30 to 60-minute intravenous infusion of KZR-261 via a central line on Days 1, 8, and 15 of a 4-week (28-day) treatment cycle.
  Up to approximately 50 participants were to be enrolled and treated with KZR-261 in Part 1 (Dose Escalation). In Part 2A (Dose Expansion), up to 175 participants (15-35 per tumor cohort [melanoma, uveal melanoma, colorectal cancer, castration-resistant prostate cancer, mesothelioma, and "All-Tumor"]) were to be enrolled. In Part 2B (Dose Optimization), up to 120 participants from up to 4 tumor types from the Dose Expansion were to be enrolled.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KZR-261 with standard therapy: open-label (Experimental): Part 1 (Dose Escalation):
  The initial dose cohort of the Dose Escalation received 1.8 mg/m2 of KZR-261. Participants received 3 doses in a 28-day cycle as an intravenous (IV) infusion for up to 6 cycles.
  _________________
  Part 2A (Dose Expansion):
  Following safety review of all Dose Escalation cohorts and determination of the maximum tolerated dose (MTD) or maximum administered dose (MAD), KZR-261 was to be evaluated for safety and preliminary efficacy in 4 tumor-specific cohorts and 1 all-tumor cohort to determine the recommended phase 2 dose (RP2D). The 4 tumor-specific cohorts will include:
  * melanoma (including uveal melanoma)
  * colorectal cancer
  * castration-resistant prostate cancer
  * mesothelioma
  Part 2B (Dose Optimization):
  Dose optimization in tumor-specific cohorts could have been initiated based on the totality of data after the MTD/MAD had been determined. Participants were to receive KZR-261 at the MTD/MAD or a lower clinically active dose of KZR-261.
  Interventions: Drug: KZR-261

INTERVENTIONS:
Drug: KZR-261 — KZR-261 for Injection is a lyophilized drug product supplied in single-use vials delivering 75 mg of KZR-261.
  Other Names: KZR-261 for Injection

SUMMARY:
A first-in-human, open-label, multicenter, Phase 1 study of KZR-261 designed to assess the safety and tolerability, preliminary anti-tumor activity, and pharmacokinetics (PK) of KZR-261, as well as identify the recommended Phase 2 dose (RP2D). The study comprised a Part 1 (Dose Escalation) and a Part 2 (2A Dose Expansion and 2B Dose Optimization) in solid organ tumors (melanoma/uveal melanoma, mesothelioma, colorectal cancer, castration-resistant prostate cancer, and "All-Tumors").

DETAILED DESCRIPTION:
The first-in-human, open-label, multicenter, Phase 1 study of KZR-261, Study KZR-261-101, was conducted in two parts (dose escalation and dose expansion) to evaluate the safety and tolerability, pharmacokinetics, pharmacodynamics, and evaluate the preliminary anti-tumor activity of KZR-261 in participants with locally advanced or metastatic solid malignancies for whom no therapeutics are available (or available therapeutics were refused) that can confer a reasonable likelihood of clinical benefit. The 5 tumor cohorts in the dose expansion part include advanced malignant:

* melanoma/uveal melanoma
* mesothelioma
* colorectal cancer
* castration-resistant prostate cancer
* "All-Tumors" (other advanced solid malignancies)

Part 1 (Dose Escalation) and Part 2 (2A Dose Expansion and 2B Dose Optimization) comprised a 4-week Screening Period, a Treatment Period lasting approximately 24 weeks, 4-6-week Safety Follow-up, and a 12-month Long-Term Follow-up Period (after last dose of study treatment), for a total study duration of approximately 20 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic evidence of malignant solid tumor with advanced disease (except primary central nervous system [CNS] neoplasms), defined as cancer that is either metastatic or locally advanced and unresectable (and for which additional radiation therapy or other locoregional therapies are not considered to result in reasonable clinical benefit).
* Disease that is resistant to or relapsed following available standard systemic therapy, or for which there is no standard systemic therapy or reasonable therapy in the Investigator's judgement likely to result in clinical benefit, or if such therapy has been refused by the subject. Documentation of the reason must be provided for subjects who have not received a standard therapy likely to result in clinical benefit.
* Eastern Cooperative Oncology Group Performance Status score of 0 or 1.
* Adequate baseline hematologic and organ function.
* Willing to use contraception.

Additional Inclusion for Part 2: Histologic or cytologic evidence of malignancy (melanoma/uveal melanoma, colorectal cancer, castration-resistant prostate cancer, mesothelioma).

Exclusion Criteria:

* Subjects who have participated in Part 1 dose escalation are not eligible to enroll in Part 2 dose expansion.
* Persistent clinically significant toxicities from previous anticancer therapy (excluding alopecia).
* Treatment with cytotoxic, biologic, or targeted therapies for advanced cancer within 14 days before administration of the subject's first dose of KZR-261.
* Treatment with an investigational drug within 28 days before administration of the subject's first dose of KZR-261.
* Radiation therapy within 14 days of before administration of the subject's first dose of KZR-261.
* Major surgical procedure within 28 days before administration of the subject's first dose of KZR-261.
* History of risk factors for Torsades de pointes.
* Active, symptomatic CNS metastases or primary CNS malignancy.
* Any female who is breastfeeding or who plans to become pregnant during the study, or who are actively trying to conceive at the time of signing of the informed consent form (ICF).
* Uncontrolled, clinically significant pulmonary disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kezar Study Director, Study Director — Kezar Life Sciences, Inc.
Locations (12):
- United States (12):
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Henry Ford Health System, Detroit, Michigan
  - University Hospitals - Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sara Cannon Research Institution (SCRI) - Tennessee Oncology Nashville, Nashville, Tennessee
  - START (South Texas Accelerated Research Therapeutics), San Antonio, Texas
  - Virginia Cancer Specialists (VCS), Fairfax, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington

REFERENCES:
- See also: Kezar Life Sciences, Inc. corporate website — http://www.kezarlifesciences.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At the time of study termination, Part 2A of the study had only enrolled participants with melanomas. Part 2B of the study (Dose Optimization) did not occur.
Groups:
- Dose 1: Participants received 1.8 mg/m^2 of KZR-261. Participants received 3 doses in a 28-day cycle as an intravenous (IV) infusion for up to six cycles.
- Dose 2: Participants received 3.6 mg/m^2 of KZR-261. Participants received 3 doses in a 28-day cycle as an intravenous (IV) infusion for up to six cycles.
- Dose 3: Participants received 7.2 mg/m^2 of KZR-261. Participants received 3 doses in a 28-day cycle as an intravenous (IV) infusion for up to six cycles.
- Dose 4: Participants received 12 mg/m^2 of KZR-261. Participants received 3 doses in a 28-day cycle as an intravenous (IV) infusion for up to six cycles.
- Dose 5: Participants received 18 mg/m^2 of KZR-261. Participants received 3 doses in a 28-day cycle as an intravenous (IV) infusion for up to six cycles.
- Dose 6: Participants received 27 mg/m^2 of KZR-261. Participants received 3 doses in a 28-day cycle as an intravenous (IV) infusion for up to six cycles.
- Dose 7: Participants received 40 mg/m^2 of KZR-261. Participants received 3 doses in a 28-day cycle as an intravenous (IV) infusion for up to six cycles.
- Dose 8; Melanoma Expansion Cohort: Participants received 60 mg/m^2 of KZR-261. Participants received 3 doses in a 28-day cycle as an intravenous (IV) infusion for up to six cycles.
- Dose 9: Participants received 80 mg/m^2 of KZR-261. Participants received 3 doses in a 28-day cycle as an intravenous (IV) infusion for up to six cycles.
Period: Overall Study
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Melanoma Expansion Cohort
Started | 2 | 2 | 2 | 6 | 6 | 6 | 5 | 17 | 8 | 7
Completed | 1 | 0 | 1 | 0 | 1 | 3 | 1 | 0 | 0 | 0
Not Completed | 1 | 2 | 1 | 6 | 5 | 3 | 4 | 17 | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Melanoma Expansion Cohort | Total
Number analyzed (Participants) | 2 | 2 | 2 | 6 | 6 | 6 | 5 | 17 | 8 | 7 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.4 (8.5) | 61.1 (3.6) | 81.4 (9.6) | 59.8 (13.2) | 67.2 (5.0) | 67.3 (6.4) | 64.4 (7.0) | 67.4 (8.8) | 59.0 (12.5) | 71.3 (10.5) | 66.0 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 4 | 3 | 5 | 5 | 8 | 5 | 4 | 34
  Male | 2 | 2 | 2 | 2 | 3 | 1 | 0 | 9 | 3 | 3 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 8
  Not Hispanic or Latino | 0 | 1 | 2 | 5 | 5 | 5 | 5 | 15 | 7 | 7 | 52
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 5
  White | 2 | 1 | 2 | 4 | 5 | 4 | 5 | 14 | 6 | 7 | 50
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 3
ECOG Performance Status at Screening [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is a scale from 0-4 used to understand patient with cancer's general well-being and function, where higher scores represent lower well-being and more limited function.
  Participants
    Zero | 1 | 0 | 1 | 0 | 1 | 2 | 4 | 3 | 3 | 4 | 19
    One | 1 | 2 | 1 | 6 | 5 | 4 | 1 | 14 | 5 | 3 | 42
    Two | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Three | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Four | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Not Done | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Type of Cancer Under Study [Count of Participants; unit: Participants]
  Breast | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Cervical | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Colorectal | 1 | 1 | 0 | 3 | 4 | 2 | 1 | 1 | 2 | 0 | 15
  Esophagus | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Gastric | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 4
  Head and Neck | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
  Lung | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 6
  Malignant Cutaneous Melanoma | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 5 | 7
  Malignant Uveal Melanoma | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3
  Mesothelioma | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Ovarian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Pancreatic | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 6 | 0 | 0 | 8
  Prostate | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Other | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 4 | 1 | 0 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Participants Experiencing Adverse Events as Assessed by CTCAE v5.0 (Part 1 & 2)
Description: Incidence and percentage of adverse events and serious adverse events will be collected from start of enrollment
Time Frame: 20 months
Population: All participants who received at least 1 dose of study treatment (KZR-261).
Measure: Number; unit: participants
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Melanoma Expansion Cohort
Number analyzed (Participants) | 2 | 2 | 2 | 6 | 6 | 6 | 5 | 17 | 8 | 7
participants
  Mild (Grade 1) | 2 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
  Moderate (Grade 2) | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 2
  Severe (Grade 3) | 0 | 0 | 0 | 3 | 4 | 4 | 1 | 5 | 2 | 0
  Life-threatening (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 12 | 5 | 5
  Death (Grade 5) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number and Percentage of Participants Experiencing Dose-limiting Toxicities
Description: Number and percentage of participants experiencing dose-limiting toxicities (DLT) collected from start of enrollment through the first 28 days of Cycle 1 as assessed by CTCAE v5.0 (Part 1).
Time Frame: 28 days
Population: The DLT Evaluable Population consists of all participants who either met the following minimal exposure criteria and have sufficient safety evaluations without having a DLT, or have experienced a DLT during the DLT assessment period. Participants who did not experience a DLT in Dose Escalation must have received all of their scheduled doses (Days 1, 8, and 15) during the DLT assessment period with completed follow-up data available through 28 days of Cycle 1 to be DLT-assessable.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9
Number analyzed (Participants) | 2 | 2 | 2 | 5 | 6 | 5 | 5 | 14 | 5
Participants | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1

3. Primary Outcome: Maximum Plasma Concentration of KZR-261 (Part 1)
Description: This is the maximum observed plasma concentration (Cmax) observed after administration of KZR-261 in Cycle 1 (Days 1 and 15) and Cycle 2 (Days 1 and 15). The PK parameters were calculated using all timepoints at which the concentration was measured, ie. predose, 15 minutes post start of infusion, end of infusion, and 5, 15, 30 minutes, 1, 2, 4, 6, 24, 48, and 96 hours post infusion.
Time Frame: Cycle 1: Day 1, Cycle 1: Day 15, Cycle 2: Day 1, and Cycle 2: Day 15
Population: The PK analyses were performed for all subjects in the PK population (all subjects that received at least one dose plasma KZR-261 concentration measurement during Cycles 1 and 2 of treatment).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Dose 1: Participants received 1.8 mg/m^2 of KZR-261.
- Dose 2: Participants received 3.6 mg/m^2 of KZR-261.
- Dose 3: Participants received 7.2 mg/m^2 of KZR-261.
- Dose 4: Participants received 12 mg/m^2 of KZR-261.
- Dose 5: Participants received 18 mg/m^2 of KZR-261.
- Dose 6: Participants received 27 mg/m^2 of KZR-261.
- Dose 7: Participants received 40 mg/m^2 of KZR-261.
- Dose 8: Participants received 60 mg/m^2 of KZR-261.
- Dose 9: Participants received 80 mg/m^2 of KZR-261.
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9
Number analyzed (Participants) | 2 | 2 | 2 | 5 | 6 | 6 | 5 | 17 | 8
ng/mL
  Cycle 1, Day 1 | 601.5 (26.9) | 1414.9 (1.5) | 1536.1 (34.7) | 2793.5 (44.9) | 5126.6 (37.8) | 7475.8 (10.9) | 9531.2 (39.5) | 12159.8 (27.8) | 16346.5 (27.4)
  Cycle 1, Day 15: number analyzed (Participants) | 2 | 1 | 2 | 5 | 5 | 6 | 5 | 15 | 5
  Cycle 1, Day 15 | 580.6 (35.5) | 2160.0 (NA) — The measure was only collected for one participant. | 2413.2 (46.0) | 4149.8 (45.6) | 4409.6 (40.2) | 7571.7 (23.8) | 11906.8 (23.6) | 12917.1 (36.0) | 25955.5 (154.2)
  Cycle 2, Day 1: number analyzed (Participants) | 2 | 2 | 2 | 3 | 5 | 4 | 4 | 10 | 3
  Cycle 2, Day 1 | 566.5 (13.3) | 1724.4 (46.7) | 2406.6 (57.4) | 3712.8 (54.5) | 4359.1 (18.7) | 6686.2 (21.1) | 14497.6 (42.2) | 12208.5 (36.0) | 31491.0 (260.2)
  Cycle 2, Day 15: number analyzed (Participants) | 2 | 2 | 2 | 2 | 4 | 4 | 4 | 5 | 1
  Cycle 2, Day 15 | 603.2 (20.7) | 1334.6 (61.3) | 2128.8 (36.3) | 3510.7 (27.5) | 4409.6 (28.6) | 7343.5 (24.9) | 12218.5 (11.0) | 15342.7 (31.4) | 18300.0 (NA) — The measure was only collected for one participant.

4. Primary Outcome: The Plasma Concentration Time Curve of KZR-261 (Part 1)
Description: This is the area under the curve (AUC) from predose through postdose observed after administration of KZR-261 in Cycle 1 (Days 1 and 15) and Cycle 2 (Days 1 and 15). The PK parameters were calculated using all timepoints at which the concentration was measured, ie. predose, 15 minutes post start of infusion, end of infusion, and 5, 15, 30 minutes, 1, 2, 4, 6, and 24 hours post infusion.
Time Frame: Cycle 1: Day 1, Cycle 1: Day 15, Cycle 2: Day 1, and Cycle 2: Day 15
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9
Number analyzed (Participants) | 2 | 2 | 2 | 5 | 6 | 6 | 5 | 17 | 8
hr*ng/mL
  Cycle 1, Day 1 | 653.2 (14.5) | 1483.4 (101.6) | 2252.7 (13.7) | 5592.0 (74.6) | 6427.1 (30.8) | 9919.2 (11.1) | 15766.7 (15.3) | 22918.9 (45.4) | 34948.3 (31.7)
  Cycle 1, Day 15: number analyzed (Participants) | 2 | 1 | 2 | 5 | 5 | 6 | 5 | 15 | 5
  Cycle 1, Day 15 | 528.6 (20.5) | 2596.4 (NA) — Only one participant had measurements at this timepoint. | 2511.2 (42.4) | 4259.1 (26.4) | 6280.1 (31.8) | 8944.0 (16.4) | 14624.8 (13.9) | 18088.1 (27.0) | 38084.6 (96.2)
  Cycle 2, Day 1: number analyzed (Participants) | 2 | 2 | 2 | 3 | 5 | 4 | 4 | 10 | 3
  Cycle 2, Day 1 | 532.2 (2.9) | 1506.8 (68.2) | 2485.0 (12.1) | 6536.5 (80.4) | 7030.0 (21.6) | 10171.0 (18.0) | 20581.5 (36.2) | 20847.3 (57.6) | 48172.7 (92.3)
  Cycle 2, Day 15: number analyzed (Participants) | 2 | 2 | 2 | 2 | 4 | 4 | 4 | 5 | 1
  Cycle 2, Day 15 | 568.6 (21.8) | 1304.5 (78.3) | 2126.4 (22.7) | 5135.9 (53.6) | 6246.6 (28.2) | 8958.0 (23.2) | 17093.8 (16.0) | 22390.0 (31.7) | 37991.6 (NA) — Only one participant had measurements at this timepoint.

5. Secondary Outcome: Objective Response (ORR) Following KZR-261
Description: The objective response following KZR-261 defined as a best overall response of Complete Response (CR) or Partial Response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. A CR is defined as the disappearance of all target lesions and a PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of longest lesion diameters.
Time Frame: 20 months
Population: The Response Evaluable Population is defined as all participants who received at least 1 dose of study treatment (KZR-261) and who have a baseline and at least 1 post-baseline anti-tumor response assessment.
Measure: Number; unit: participants
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Melanoma Expansion Cohort
Number analyzed (Participants) | 2 | 2 | 2 | 5 | 4 | 5 | 5 | 14 | 6 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Participants With Clinical Benefit of Stable Disease Following KZR-261
Description: The clinical benefit rate defined as the number of participants achieving a best response of complete response (CR)/partial response (PR) or stable disease over at least 2 consecutive response assessment time points. Stable disease is defined as neither sufficient decrease to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum of longest diameters of target lesions while on study.
Time Frame: 20 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Melanoma Expansion Cohort
Number analyzed (Participants) | 2 | 2 | 2 | 5 | 4 | 5 | 5 | 14 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 0 | 1

7. Secondary Outcome: Progression-free Survival of Participants Treated With KZR-261
Description: The number of participants with progression-free survival (PFS), defined as the date of initiation of study treatment to the date of documented PD or death from any cause, whichever occurs first, at 4 months and 6 months. PFS is based on the number of subjects in each group in the response evaluable population at the specific timepoints (4 or 6 months).
Time Frame: 4 months and 6 months
Population: The Response Evaluable Population is defined as all subjects who receive at least 1 dose of study treatment (KZR-261) and who have a baseline and at least 1 post-baseline anti-tumor response assessment. For participants who have neither progressed nor died, PFS is censored at the date of the last disease assessment. PFS at 4 months and 6 months are defined as subjects alive and progression-free at 4 months and at 6 months, respectively, after the initiation of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Melanoma Expansion Cohort
Number analyzed (Participants) | 2 | 2 | 2 | 5 | 4 | 5 | 5 | 14 | 6 | 6
Participants
  4 Months: number analyzed (Participants) | 2 | 2 | 2 | 5 | 4 | 4 | 5 | 14 | 6 | 6
  4 Months | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 0 | 1
  6 Months: number analyzed (Participants) | 2 | 2 | 2 | 5 | 4 | 3 | 5 | 14 | 6 | 6
  6 Months | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1

8. Secondary Outcome: Overall Survival of Participants Treated With KZR-261
Description: Time of overall survival for participants treated with KZR-261.
Time Frame: 20 months
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Melanoma Expansion Cohort
Number analyzed (Participants) | 2 | 2 | 1 | 5 | 1 | 2 | 2 | 10 | 2 | 4
weeks | 21.7 [21.0 to NA] — NA = Not calculable because the event of interest did not occur in a sufficient number of participants to allow estimation. | 22.6 [12.6 to NA] — NA = Not calculable because the event of interest did not occur in a sufficient number of participants to allow estimation. | NA [15.0 to NA] — NA = Not calculable because the event of interest did not occur in a sufficient number of participants to allow estimation. | 17.9 [8.4 to NA] — NA = Not calculable because the event of interest did not occur in a sufficient number of participants to allow estimation. | NA [39.7 to NA] — NA = Not calculable because the event of interest did not occur in a sufficient number of participants to allow estimation. | NA [33.9 to NA] — NA = Not calculable because the event of interest did not occur in a sufficient number of participants to allow estimation. | 53.4 [11.7 to NA] — NA = Not calculable because the event of interest did not occur in a sufficient number of participants to allow estimation. | 12.4 [7.9 to 26.1] | NA [9.3 to NA] — NA = Not calculable because the event of interest did not occur in a sufficient number of participants to allow estimation. | 24.6 [19.4 to NA] — NA = Not calculable because the event of interest did not occur in a sufficient number of participants to allow estimation.

ADVERSE EVENTS:
Time Frame: Through end of study, up to 2.25 years
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 | Dose 7 | Dose 8 | Dose 9 | Melanoma Expansion Cohort
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 1/6 | 1/6 | 0/6 | 0/5 | 0/17 | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 3/6 | 3/6 | 3/6 | 0/5 | 8/17 | 4/8 | 4/7
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 1/2 | 6/6 | 6/6 | 6/6 | 5/5 | 17/17 | 7/8 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose 1 (N=2) | Dose 2 (N=2) | Dose 3 (N=2) | Dose 4 (N=6) | Dose 5 (N=6) | Dose 6 (N=6) | Dose 7 (N=5) | Dose 8 (N=17) | Dose 9 (N=8) | Melanoma Expansion Cohort (N=7)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders and administration site conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders and administration site conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose 1 (N=2) | Dose 2 (N=2) | Dose 3 (N=2) | Dose 4 (N=6) | Dose 5 (N=6) | Dose 6 (N=6) | Dose 7 (N=5) | Dose 8 (N=17) | Dose 9 (N=8) | Melanoma Expansion Cohort (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 5 (9) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 6 (15) | 1 (1) | 2 (6)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract nuclear (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 1 (2) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (6) | 3 (5) | 2 (4) | 5 (5) | 1 (2) | 4 (5)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Salivary gland pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 6 (6) | 2 (2) | 4 (5)
Asthenia (General disorders and administration site conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site rash (General disorders and administration site conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders and administration site conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Face oedema (General disorders and administration site conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders and administration site conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 5 (8) | 3 (4) | 1 (1)
Gait disturbance (General disorders and administration site conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised oedema (General disorders and administration site conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders and administration site conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Nodule (General disorders and administration site conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders and administration site conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders and administration site conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Peripheral swelling (General disorders and administration site conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders and administration site conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (26) | 10 (28) | 3 (6) | 3 (11)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (31) | 2 (10) | 0 (0) | 2 (6)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejaculation disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Penile oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 4 (4) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/36/NCT05047536/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT05047536/SAP_001.pdf